CLINICAL TRIAL: NCT04032717
Title: A Randomized, Double-Blind Phase 1 Safety and Pharmacokinetic Study of Q-Griffithsin Enema Administered Rectally to HIV-1 Seronegative Adults
Brief Title: Griffithsin-based Rectal Microbicide for PREvention of Viral ENTry (PREVENT)
Acronym: PREVENT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, study enrollment has been prematurely terminated.
Sponsor: Rhonda Brand (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Intrucept Biomedicine LLC (Unknown)
Responsible Party: Sponsor-Investigator, Rhonda Brand, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY19030322; U19AI113182 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-07-25 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: HIV Prevention
Keywords: microbicide; enema; receptive anal intercourse; HIV prevention; HIV transmission
MeSH Terms: interventions — q-griffithsin; Enema

STUDY DESIGN:
Intervention Model Description: randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Arm 1 will enroll 3 participants to receive the open-label Q-GRFT enema. The remaining 18 participants will be randomized 2:1 (Q-GRFT enema: placebo enema) resulting in twelve participants enrolled into Arm 2 and six participants enrolled into Arm 3. The randomization scheme will be generated by the statistical group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-label Q-GRFT enema (Experimental): Open-label Q-GRFT enema administered rectally once as a single dose (Arm 1)
  Interventions: Drug: Q-Griffithsin (Q-GRFT) enema
- Randomized, blinded Q-GRFT enema (Experimental): Blinded Q-GRFT enema administered rectally once as a single dose (Arm 2)
  Interventions: Drug: Q-Griffithsin (Q-GRFT) enema
- Randomized, blinded placebo enema (Placebo Comparator): Blinded placebo enema administered once as a single dose (Arm 3)
  Interventions: Other: Placebo enema

INTERVENTIONS:
Drug: Q-Griffithsin (Q-GRFT) enema — Investigational enema composed of 4.2mL Q-Griffithsin (Q-GRFT) 9.6mg/mL combined with approximately 120.8mL of 0.9% sodium chloride solution to yield an active enema study product that will contain and deliver a dose of approximately 40mg of Q-GRFT
  Other Names: Study product enema
  Arms: Open-label Q-GRFT enema; Randomized, blinded Q-GRFT enema
Other: Placebo enema — Approximately 125mL of 0.9% sodium chloride solution
  Arms: Randomized, blinded placebo enema

SUMMARY:
This is the first-in-human clinical study to see if a single dose of an investigational enema made from a modified plant protein called Q-Griffithsin is safe, tolerated, and acceptable for use by healthy adults 18-45 years of age who practice receptive anal intercourse.

DETAILED DESCRIPTION:
A microbicide is a drug or agent designed to prevent transmission of HIV. Griffithsin, or "GRFT", is an investigational product that is being developed as a microbicide. GRFT is a naturally occurring protein originally isolated from the red alga Griffithsia found in the South Pacific Ocean. GRFT is one of the most powerful, broad-spectrum antivirals ever tested and its activity is under study for potential therapeutic applications against several viral pathogens including HIV, herpes simplex virus type-2, human papillomavirus (HPV), and hepatitis C. GRFT can be formulated into a number of delivery vehicles including gels, films, suppositories and even simple enemas or rinses.

The product is intended for use prior to sexual activity by people who practice receptive anal intercourse (RAI), and thus represent the population most vulnerable to HIV-1 transmission due to the high concentration of HIV target cells in the rectal mucosa and the presence of mucosal trauma commonly associated with RAI. For the purposes of this study GRFT has been genetically modified to produce a more stable compound less prone to oxidation, Q-GRFT.

Up to 21 HIV-uninfected individuals between the ages of 18 - 45 years will be enrolled in this study at the University of Pittsburgh, the only study site. Participants will be screened to exclude those with HIV infection, and anorectal sexually transmitted infections (STIs) (Visit 1). Up to 28 days after screening, eligible participants will return for a baseline visit (Visit 2), be assigned to a study arm, and undergo sample collection including flexible sigmoidoscopy with collection of colorectal biopsies.

The first 3 participants will be assigned to Arm 1 and receive a clinician administered single dose exposure of open-label Q-GRFT. Once the participants in Arm 1 complete Visit 4, study activity will be paused while the study Protocol Safety Review Team (PSRT) conducts an interim review of the clinical and laboratory data. In the absence of any significant safety concerns, the PSRT will be asked to approve enrollment of Study Arms 2 and 3. The remaining 18 participants will be assigned 2:1 in a randomized and blinded fashion to either Study Arm 2 (Q-GRFT) or 3 (placebo), respectively.

At Visit 3, participants will receive a clinician-administered single-dose exposure followed by flexible sigmoidoscopy with collection of colorectal biopsies at 1-hr and PK sampling of blood and rectal fluid at 1-hr and 4-hr. Participants will return to clinic the next day (Visit 4) for colorectal biopsies and 24-hr PK sampling. Participants in Arm 1 will additionally return for PK sampling including colorectal biopsies at 48 hrs (Visit 4a) following Visit 3. Participants will be contacted by study staff approximately 3 days after Visit 4 to collect safety information.

Participants will return for a final study visit, Visit 5, 4 weeks +/- 1 week after Visit 4/4a to collect blood samples for PK and immunogenicity assessments. A final study exit call for safety will occur within one week after the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 45 years at screening, verified per site SOP
2. Male participants, born male; female participants, born female.
3. Availability to return for all study visits, barring unforeseen circumstances
4. Willing and able to

   * communicate in English
   * provide written informed consent to take part in the study
   * provide adequate locator information, as defined in site SOP
5. Must agree

   * not to participate in other concurrent interventional and/or drug trials
   * to use study-provided condoms for vaginal or anal intercourse for the duration of the study
   * to avoid insertion of anything in the vagina or rectum (e.g., penis, sex toy, medication, enemas) 72 hours before and after study product exposure and rectal sampling visits
6. Understands and agrees to local STI reporting requirements
7. HIV-1 seronegative at screening and enrollment
8. A history of RAI at least 5 times in lifetime and once in the prior year. (Required to assure that participants are comfortable with study procedures and study product administration.)
9. Must be in general good health in the opinion of the investigator
10. Using an effective method of contraception and intending to continue use of an effective method for the duration of study participation. Acceptable methods include:

    1. Males

       * male condoms
       * sterilization of participant or partner
       * partner use of hormonal contraception or intrauterine device [IUD]
       * identifies as a man who has sex with men exclusively
       * and/or sexually abstinent for the past 90 days
    2. Females

       * hormonal methods
       * IUD inserted at least 28 days prior to enrollment
       * sterilization of participant or partner
       * and/or sexually abstinent for the past 90 days

    In addition to the criteria listed above, female participants must meet the following criteria:
11. Not pregnant or breastfeeding
12. Regular menstrual cycles of approximately 21 to 35 days apart with no untreated intermenstrual bleeding

Note: This criterion is not applicable to participants using continuous combination oral contraceptive pills or progestin-only methods (such as Depo-Provera or levonorgestrel-releasing IUD), as the absence of regular menstrual cycles is an expected, normal consequence in this context.

Exclusion Criteria:

1. Undergoing or completed gender reassignment
2. Participant reports any of the following at Screening:

   1. Post-exposure prophylaxis for HIV exposure within 4 weeks prior to screening
   2. Condomless insertive or receptive anal intercourse with more than one partner in the past six months
   3. Known HIV-positive sexual partner within the last 6 months
   4. History of STI in the last 3 months
   5. Transactional sex within the last 12 months
   6. Non-therapeutic injection drug use in the 12 months prior to screening
   7. Any use of methamphetamine, gamma hydroxybutyrate, cocaine or heroin in the 12 months prior to screening
   8. History of recurrent urticaria
   9. Use of antiretroviral medications with activity against HIV within the 4 weeks prior to the Enrollment, including PrEP with Truvada®
   10. Use of systemic immunomodulatory medications within the 4 weeks prior to the Enrollment
   11. Use of rectally administered medications or products (including condoms) containing Nonoxynol-9 (N-9) within the 4 weeks prior to the Enrollment
   12. Participating in another research study involving drugs or medical devices within the 4 weeks prior to the Enrollment
   13. Has plans to relocate away from the study site area during the period of study participation
3. Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation:

   1. Heparin, including Lovenox® (enoxaparin sodium)
   2. Warfarin
   3. Plavix® (clopidogrel bisulfate)
   4. Any other drugs that are associated with increased likelihood of bleeding following mucosal biopsy (e.g., daily high dose aspirin > than 81 mg, NSAIDs, or Pradaxa®)
   5. Rectally or vaginally administered medications (including over-the-counter products)
   6. Antiretroviral medications with activity against HIV
4. History of significant gastrointestinal bleeding in the opinion of the investigator
5. Abnormalities of the colorectal mucosa, or significant symptom(s), which in the opinion of the clinician represents a contraindication to protocol-required biopsies (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids).
6. At screening: participant-reported symptoms, and/or clinical or laboratory diagnosis of active rectal or reproductive tract infection requiring treatment per current CDC guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include CT, GC, syphilis, active HSV lesions, chancroid, genital sores or ulcers, or symptomatic genital warts requiring treatment.

   Note:

   • HSV-1 or HSV-2 seropositive diagnosis with no active lesions is allowed, since treatment is not required
7. Has any of the following laboratory abnormalities at Screening:

   1. White blood cell count Grade 2 or higher
   2. Hemoglobin Grade 1 or higher
   3. Platelet count Grade 1 or higher
   4. International Normalized Ratio (INR) Grade 2 or higher
   5. Calculated creatinine clearance ≤ 70 mL/minute using the Cockcroft-Gault equation:

      ♀: (140 - age in yrs) x (weight in kg) x (0.85)/72 x (serum Cr in mg/dL)

      ♂: (140 - age in yrs) x (weight in kg) /72 x (serum Cr in mg/dL)
   6. Grade 2 or higher ALT and/or AST
   7. Grade 2 or higher Total bilirubin
   8. Positive for Hepatitis B surface antigen (HBsAg)
   9. Positive for Hepatitis C antibody (HCV Ab)
   10. Positive for HIV
8. Any other condition or prior therapy that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, current or recent history of severe, progressive, or uncontrolled substance abuse, or renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease

   In addition to the criteria listed above, female participants will be excluded if they meet any of the following criteria:
9. Participant reports any of the following at Screening:

   1. Last pregnancy outcome or gynecological surgery 90 days or less prior to screening
   2. Intends to become pregnant during the period of study participation
   3. Chronic and/or recurrent symptomatic vaginal candidiasis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will exclude transgender populations. Although it is recognized that this is a critical group to include in the evaluation of new HIV prevention products it is felt that inclusion of transgender populations would increase the heterogeneity of the study population and it is not clear what the impact of exogenous hormones might be on immunological or pharmacokinetic parameters being evaluated in the study.
Enrollment: 18 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
The number and frequency of adverse events Grade 2 or higher and genitourinary adverse events Grade 1 or higher | Baseline through the final study contact, or about 8 weeks
  Safety analysis will be conducted on all participants who have receive study product. The number and the frequency of ≥ Grade 2 adverse events (AEs) and ≥ Grade 1 Genitourinary AEs as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric AEs, Version 2.1 (March 2017), Addendum 1 Female Genital Grading Table for Use in Microbicide Studies (November 2007), and/or Addendum 3 Rectal Grading Table for Use in Microbicide Studies (Clarification dated May 2012) to this table will be tabulated for each of the three methods of administration from Baseline through the final study contact. To determine whether AEs are occurring excessively, the proportion of subjects that experience an AE will be calculated for each method of administration. Additional safety analyses will also tabulate the number and type of AEs observed overall, and by severity, site, and study product. AEs that lead to discontinuation of study participation will be tabulated separately.
The proportion of participants who report product characteristics to be considered a barrier in study product use, operationalized as having a rating of lower than 3 on a 5-point Likert scale, in disliking or likelihood of future use | Once 24 hours post-dose
  One day after study product administration, participants will complete an acceptability questionnaire to provide descriptive statistics on participants' opinions on the enema's characteristics, application process, the applicator design and the use-regimen, as well as the degree to which participants believe these characteristics and side-effects could pose barriers in future sustained use. On a 5-point Likert scale, with 1 being completely unacceptable and 5 being highly acceptable, the distributions of scores on all product characteristics will be examined to determine product characteristics that pose or could pose significant barriers in current or future product use.
Area under the concentration-time curve (AUC) of Q-GRFT | Pre-dose and 1, 4, and 24 hours post-dose
  AUC of Q-GRFT as measured in plasma, rectal fluid, rectal mucosal tissue homogenates, and enema fluid effluent.
Maximum concentration (Cmax) of Q-GRFT | Pre-dose and 1, 4, and 24 hours post-dose
  Cmax of Q-GRFT as measured in plasma, rectal fluid, rectal mucosal tissue homogenates, and enema fluid effluent.
Time to maximum concentration (Tmax) of Q-GRFT | Pre-dose and 1, 4, and 24 hours post-dose
  Tmax of Q-GRFT as measured in plasma, rectal fluid, rectal mucosal tissue homogenates, and enema fluid effluent .
Minimum concentration (Cmin) of Q-GRFT | Pre-dose and 1, 4, and 24 hours post-dose
  Cmin of Q-GRFT as measured in plasma, rectal fluid, rectal mucosal tissue homogenates, and enema fluid effluent.
Half-life (t½) of Q-GRFT | Pre-dose and 1, 4, and 24 hours post-dose
  t½ of Q-GRFT as measured in plasma, rectal fluid, rectal mucosal tissue homogenates, and enema fluid effluent.

SECONDARY OUTCOMES:
Change in humoral antibody responses to Q-GRFT in blood by ELISA and PBMC Q-GRFT antigen stimulation | Baseline and 4 weeks post-dose
  The titer of immunoglobulins in blood and rectal secretions will be assessed. Lymphocytes collected from peripheral blood will be stimulated with Q-GRFT and an ELISPot assay used to quantify number of B-cells that produce specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Ho, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- HIV/AIDS Clinical Research Unit / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The awardee institution will follow Federal grant policies concerning the sharing of research data. The awardee institution will share its information, data and resources among its own researchers and the collaborating researchers as well as with researchers at other institutions. The research team will make the results of this collaboration and any accompanying data available to the public. In accordance with Federal policies on Data Sharing, research data will be made available to researchers and/or the general public as requested. The limitations on this policy are that data will not generally be available until such a time that it is submitted for publication. Also, all human subjects' rights to privacy with respect to any human tissue samples to be used as a part of this study will be approved by the appropriate regulatory boards, protected and de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication

REFERENCES:
- [Derived] Shrivastava-Ranjan P, Lo MK, Chatterjee P, Flint M, Nichol ST, Montgomery JM, O'Keefe BR, Spiropoulou CF. Hantavirus Infection Is Inhibited by Griffithsin in Cell Culture. Front Cell Infect Microbiol. 2020 Nov 4;10:561502. doi: 10.3389/fcimb.2020.561502. eCollection 2020. PMID 33251157

DOCUMENTS (1):
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04032717/ICF_000.pdf